CLINICAL TRIAL: NCT01639014
Title: Effect of 3-month Treatment With F2695 (75mg OD) on Improving Functional Recovery of Patients With Ischemic Stroke. A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-Controlled Study
Brief Title: Effect of F2695 on Functional Recovery After Ischemic Stroke
Acronym: LIFE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F02695 LP 2 05; 2012-001592-37 (EudraCT Number)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- F2695 (Experimental)
  Interventions: Drug: F2695
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: F2695 — 75 mg OD in 2 capsules
  Arms: F2695
Drug: placebo — 2 capsules
  Arms: placebo

SUMMARY:
The purpose of the study is to assess the efficacy of a new serotonin-norepinephrine reuptake inhibitor (SNRI) nin functional recovery after ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, 18 to 80 years of age
* Confirmed acute ischemic stroke within the past 2 - 10 days
* Unilateral motor deficit,
* National Institutes of Health stroke scale (NIHSS) motor score >= 5
* Modified Rankin Scale (mRS) of 4 or 5
* Able and willing to comply with the site rehabilitation program requirements

Exclusion Criteria:

* Aphasia
* Severe post-stroke condition
* Active depressive episode
* Intra-cerebral hemorrhage
* Use of anti-depressant drugs
* Cardiac rhythm disorder
* Uncontrolled arterial hypertension
* Other severe acute or chronic medical or psychiatric condition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a Modified Rankin Scale (mRS) less than or equal to 1 at Week 12 | week 12

SECONDARY OUTCOMES:
Percentage of patients with NIHSS score less than or equal to 5 at Week 12 | week 12
Percentage of patients with at least one moderate to severe depressive | Baseline to week 12
Change from baseline to Week 12 of the mean NIHSS total and motor scores | baseline to week 12
Safety and tolerability assessed by the investigator including SAEs, AEs, vital signs, ECG,physical examination and laboratory tests | baseline to week 12
Percentage of patients with a mRS score less than or equal to 2 at Week 12 | baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: François Chollet, Principal Investigator — Hôpital Purpan
Locations (87):
- Belgium (7):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuis Gasthuisberg, Leuven
  - Clinique Saint-Joseph, Liège
  - Regional Ziekenhuis Sint-Trudo, Sint-Truiden
  - Sint-Andriesziekenhuis, Tielt
  - Academisch Ziekenhuis Sint Augustinus, Wilrijk
- Czechia (6):
  - Fakultní nemocnice u sv. Anny v Brne, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Kralové
  - Litomyšlská Nemocnice, a.s., Litomyšl
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultní Nemocnice Ostrava, Ostrava
  - Vítkovická nemocnice a.s., Ostrava - Vítkovice
- France (9):
  - Hopital Jean Minjoz Centre Hospitalier Universitaire Besancon, Besançon
  - Clinique des Cèdres, Cornebarrieu
  - Centre Hospitalier de Lens, Lens
  - Hôpital Roger Salengro, Lille
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hopital Lariboisière, Paris
  - Centre Hospitalier Universitaire de Poitiers Hôpital de la Milétrie, Poitiers
  - Centre Hospitalier Universitaire de Saint Etienne, Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Purpan, Toulouse
- Germany (10):
  - Neurologische Klinik GmbH, Bad Neustadt/Saale
  - Universitätsklinik Charité, Campus Mitte, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Freiburger Universitätsklinik, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Asklepios Fachklinikum Teupitz, Teupitz
- Hungary (11):
  - Jahn Ferenc Dél-pesti Kórház, Budapest
  - Magyar Honvédség Honvédkórház, Budapest
  - Semmelweis Egyetem Neurológiai Klinika, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Kaposi Mór Megyei Oktató Kórhaz, Kaposvár
  - BAZ Megyei és Egyetemi Oktató Kórház, Miskolc
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Jósa András Oktató Kórház, Nyíregyháza
  - Soproni Erzsébet Oktató Kórház, Sopron
  - Fejér Megyei Szent György Kórház, Székesfehérvár
- Italy (6):
  - Azienda Sanitaria Ospedaliera "San Giovanni Battista", Foligno
  - Azienda Ospedaliera San Gerardo, Monza
  - IRCCS "Istituto Neurologico C. Mondino", Pavia
  - Ospedale Santa Maria della Misericordia, Perugia
  - IRCCS Fondazione Santa Lucia, Roma
  - Istituto Clinico Humanitas, Rozzano
- Portugal (5):
  - Hospital Garcia de Orta, Almada
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto / Hospital Geral de Santo António, Porto
  - Hospital de São João, Porto
- Russia (13):
  - Municipal Healthcare Institution "Municipal Clinical Hospital # 3", Chelyabinsk
  - Professor S.V. Ochapovsky Territorial Clinical Hospital #1, Krasnodar
  - Clinical Hospital Number 31, Moscow
  - Non-state Healthcare Institution "N.A. Semashko Central Clinical Hospital #2 of JSC "Russian Railway, Moscow
  - Scientific Research Neurology Institute of Russian Academy of Medical Services, Moscow
  - State Budget Healthcare Institution "City clinical hospital #20", Moscow
  - State Institution of Healthcare of Moscow City "City Clinical Hospital #61", Moscow
  - State Institution "Saint Petersburg I.I. Dzhanelidze Research Institute of Emergency", Petersburg Saint
  - Municipal Medical Institute "N.I.Pirogov City Clinical hospital #1", Samara
  - State Healthcare Institution "Samara M.I.Kalinin Regional Clinical Hospital", Samara
  - Smolensk State Medical Academy of RosZdrav, Smolensk
  - Bashkirian State Medical University, Ufa
  - Regional Hospital #1, Ekaterinburg, Yekaterinburg
- Spain (11):
  - Hospital General de Albacete, Albacete
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital de Tortosa Verge de la Cinta, Tortosa
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Sweden (6):
  - Danderyds Sjukhus AB, Danderyd
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Universitetssjukhuset Linköping, Linköping
  - Skånes Universitetssjukhus i Lund, Lund
  - Mora lasarett, Mora
  - Kärnsjukhuset i Skövde-KSS, Skövde
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Klinik Hirslanden, Zurich